CLINICAL TRIAL: NCT04721938
Title: Healthy Parents - Healthy Children. Weight Loss Before Fertility Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-048-2019
Record Dates: First submitted 2020-06-16; First posted 2021-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Infertility; Overweight and Obesity; Weight Loss; Vaginal Flora Imbalance; DNA Damage
Keywords: female infertility; male infertility; life style intervention; vaginal microbiome; synthetic endocrine disrupting chemicals; EDCs; DNA fragmentation index; DFI; gene expression
MeSH Terms: conditions — Infertility; Overweight; Obesity; Weight Loss; Infertility, Female; Infertility, Male

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Systematic weight loss intervention
  Interventions: Behavioral: Systematic weight loss intervention

INTERVENTIONS:
Behavioral: Systematic weight loss intervention — Weight reduction through life style changes in diet and exercise by the following means:
  * Counselling with a Nutritionist Nurse on diet and exercise
  * Online Smartphone coaching program (Life-sum App)
  * Motivational and adjustment dialogue and counselling with Nutritionist Nurse including anthropometric measures every month

SUMMARY:
The detrimental effect of overweight and obesity on fecundity has been well documented.

The investigators wish to investigate the intervention program for weight loss before fertility treatment.

Subsequently to gain knowledge on the effect of overweight/obesity and weight loss on the vaginal microbiome, on DNA damage on sperm cells, on the occurrence of endocrine disruptors in the endometrium, and on the gene expression in the endometrium.

DETAILED DESCRIPTION:
Purpose and aim of the study The Fertility Clinic at Zealand University Hospital wishes to introduce a new care concept: 'Healthy Parents - Healthy Children´ with the purpose of changing the behaviours of infertile men and women towards a healthier life style now and for future generations.

The Zealand Region includes areas of significant deprivation compared to Copenhagen and has a higher prevalence of obesity and poor diet.

These inequalities generate socio-demographic and long-term health challenges, decrease the chance of becoming pregnant and increase risk of life style related diseases for parents and their offspring in the long term.

The waiting time before fertility treatment (12 months in the region) represents a unique window of opportunity to encourage long-term life style changes. The aforementioned reasons initiated the planned Preconception Clinic 'Healthy Parents - Healthy Children´.

The Preconception Clinic utilises waiting list time to optimise parental health prior to conception. We will provide weight loss interventions aimed at helping the patients to a healthier lifestyle, an increased chance of conception and a decreased risk of life style diseases for themselves and their future offspring.

Purpose of study:

Patient weight loss of at least 10% at the end of intervention and at annular follow up until 5 years.

Study population: Sub-fertile population referred to the Fertility Clinic Region Zealand due to infertility.

Inclusion criteria:

20 women and 20 men with a BMI>30, age 18-40 years.

Exclusion criteria:

Inability to understand the written and oral information.

Baseline and end of intervention-sampling:

1. Blood tests (metabolic markers), blood tests for Biobank and for miRNA biomarkers
2. Urine sample
3. Women: Endometrial biopsy and vaginal swab for microbiome testing
4. Men: Sperm sample

Intervention: Weight reduction through life style changes in diet and exercise by the following means:

* Counselling with a Nutritionist Nurse on diet and exercise.
* Online smartphone coaching program (LifeSum-App)
* Motivational and adjustment dialogue and counselling with Nutritionist Nurse including anthropometric measures every month.

Primary endpoint: Weight loss of at least 10%.

Anticipated impact The aim of this study is to find a feasible intervention that can change adverse life styles in a preconception setting. Elements from the weight loss intervention can be incorporated to the broader community, for instance as Preconception weight loss packages in the local municipalities, aimed at optimizing health before conception in the general fertile population.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30
* Referred to The Fertility Clinic, Zealand Region

Exclusion Criteria:

* Unable to speak and read Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 month
  The change in weight (in kilograms) from baseline to the 6 month

SECONDARY OUTCOMES:
Change in the semen quality 1 | 6 months
  The change in the morphological semen parameters, from baseline to 6 month will be measured by using WHO recommendation for semen analysis: Sperm count (mill/ml),
Change in the semen quality 2 | 6 months
  The change in the morphological semen parameters, from baseline to 6 month will be measured by using WHO recommendation for semen analysis: Sperm concentration (ml)
Change in the semen quality 3 | 6 months
  The change in the morphological semen parameters, from baseline to 6 month will be measured by using WHO recommendation for semen analysis: Sperm motility (mill/ml)
Change in the semen quality 4 | 6 months
  The change in the morphological semen parameters, from baseline to 6 month will be measured by using WHO recommendation for semen analysis: Sperm morphology (percent)
Change in the DNA fragmentation index (DFI) | 6 months
  The change in DNA fragmentation index is measured by SPZlab using the SDI®-test
Change in the vaginal microbiome | 6 months
  The change in the vaginal microbiome will be investigated at Statens Serum Institute (SSI), measured by PCR
Change in the occurence of synthetic endocrine disruption chemicals (EDCs) | 6 month
  The change in the occurrence of synthetic endocrine disruption chemicals (EDCs) endometrium is measured by The Department of Growth and Reproduction at Rigshospitalet by using LC-MS/MS analyze
Change in MicroRNA | 6 months
  The change in MicroRNA will be measured froom blood samples and is is analysed by Department of Science and Environment, RUC
Change in the gene expression of gene involved in implantation | 6 months
  The change in the gene expression in the endometrium is analysed by Department of Science and Environment, RUC
Numbers of achieved pregnancy | Gestational week 4-8
  Both biochemical and clinical
Numbers of life births | From 9 month after inclusion
  Life birth

OTHER OUTCOMES:
Blood pressure (Systolic and Diastolic) | 6 months
Metabolic and cardiovascular marker (blood sample) 2 | 6 months
  The change in: Hemoglobin (mmol/L
Metabolic and cardiovascular marker (blood sample) 3 | 6 months
  alanine Aminotransferase (ALT)(U/L)
Metabolic and cardiovascular marker (blood sample) 4 | 6 months
  cholesterol (mmol/L)
Metabolic and cardiovascular marker (blood sample) 5 | 6 months
  triglycerides (mmol/L)
Metabolic and cardiovascular marker (blood sample) 6 | 6 months
  HbA1c (mmol/mol (IFCC)
Metabolic and cardiovascular marker (blood sample) 7 | 6 months
  creatinine (µmol/L)
Metabolic and cardiovascular marker (blood sample) 8 | 6 months
  fasting glucose level (mmol/L (eAG))

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lis Mikkelsen, MD, PhD, Study Director — The Fertility Clinic, Zealand University Hospital
Locations (1):
- The Fertility Clinic, Zealand University Hospital, Køge, Denmark